CLINICAL TRIAL: NCT01635764
Title: A Phase 3, Open-Label Study of the Safety and Efficacy of Adalimumab in Subjects With Moderate to Severe Hidradenitis Suppurativa - PIONEER (Open-Label Extension)
Brief Title: Open-label Study of the Safety and Efficacy of Adalimumab in the Treatment of Hidradenitis Suppurativa
Acronym: PIONEER (OLE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-555; 2011-003478-98 (EudraCT Number)
Record Dates: First submitted 2012-03-02; First posted 2012-07-10 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Hidradenitis Suppurativa
Keywords: hidradenitis suppurativa; open-label; acne inversa; PIONEER (OPEN-LABEL EXTENSION); adalimumab; HS; acne; tumor necrosis factor; abscess; inflammatory nodule
MeSH Terms: conditions — Hidradenitis Suppurativa; Acne Vulgaris; Abscess | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab Every Week (Experimental): Adalimumab 40 mg every week.
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — Adalimumab pre-filled syringe, administered by subcutaneous injection
  Other Names: Humira

SUMMARY:
The purpose of this study to evaluate the long term safety, tolerability and efficacy of adalimumab in subjects with moderate to severe hidradenitis suppurativa (HS).

DETAILED DESCRIPTION:
HS is a painful, chronic skin disease characterized by recurrent inflamed nodules and abscesses, which may rupture to form fistulas and subsequent scarring. This study is an open-label extension study available to subjects who participated in a prior adalimumab study who meet all the inclusion and none of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who previously participated in a prior Phase 3 AbbVie hidradenitis suppurativa (HS) study (M11-313 or M11-810) and:

  1. Completed the study; or
  2. Experienced a loss of response (LOR); or
  3. Experienced worsening or absence of improvement

     Exclusion Criteria:
* Prior treatment with any other anti-tumour necrosis factor (anti-TNF) therapy (e.g., infliximab, etanercept), or participation in an adalimumab trial other than a prior Phase 3 AbbVie HS study.
* Subject received any oral antibiotic treatment for HS within 28 days prior to the Baseline visit, except for antibiotics permitted in a prior Phase 3 AbbVie HS study.
* Subject received prescription topical therapies for the treatment of HS within 14 days prior to the Baseline visit of Study M12-555.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

REFERENCES:
- See also: Related Info. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were evaluated for entry into Study M12-555 at the final study visit of the prior phase 3 study in which they participated. Therefore, the Study M12-555 Week 0 visit and administration of the first dose of study drug in Study M12-555 was performed on the same day as the final or last visit of the prior Phase 3 study.
Period: Overall Study
Arm/Group | Adalimumab Every Week
Started | 508
Completed | 235
Not Completed | 273
Not completed — Adverse Event | 46
Not completed — Lack of Efficacy | 76
Not completed — Exceed Protocol-specified Interventions | 2
Not completed — Protocol Deviation | 1
Not completed — Withdrew Consent | 67
Not completed — Lost to Follow-up | 53
Not completed — Other | 28

BASELINE CHARACTERISTICS:
Population: Baseline characteristics provided by reporting groups defined by treatment received in the prior phase 3 studies, plus adalimumab every week (EW) received in M12-555. Baseline defined as the last measurement prior to the first dose of study drug in the prior phase 3 study (M11-810 or M11-310 for baseline characteristics.
Groups:
- EW/EW/EW: All participants who received adalimumab 40 mg every week (EW) in both Period A and Period B of the prior Phase 3 studies.
- EW/EOW/EW: All participants who received adalimumab 40 mg every week (EW) in Period A and 40 mg every other week (EOW) in Period B in the prior Phase 3 studies.
- EW/PBO/EW: All participants who received adalimumab 40 mg every week (EW) in Period A and placebo in Period B in the prior Phase 3 studies.
- PBO/EW/EW: All participants who received placebo in Period A and adalimumab 40 mg every week (EW) in Period B in prior phase 3 study M11-313.
- PBO/PBO/EW: All participants who received placebo in both Period A and Period B in prior phase 3 study M11-810.
- Total: Total of all reporting groups
Arm/Group | EW/EW/EW | EW/EOW/EW | EW/PBO/EW | PBO/EW/EW | PBO/PBO/EW | Total
Number analyzed (Participants) | 88 | 90 | 92 | 115 | 123 | 508
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (10.27) | 36.1 (10.50) | 36.5 (11.06) | 38.5 (11.92) | 37.0 (12.28) | 36.8 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 60 | 50 | 79 | 83 | 328
  Male | 32 | 30 | 42 | 36 | 40 | 180

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in the EW/EW/EW, EW/EOW/EW, and EW/PBO/EW Analysis Populations Achieving Clinical Response Per Hidradenitis Suppurativa Clinical Response (HiSCR) at Each Visit
Description: Clinical response per HiSCR defined as percent reduction from baseline of the prior phase 3 study in the abscess and inflammatory nodule ≥ 50% (AN50) with no increase in the abscess count and no increase in the draining fistula count. Last Observation Carried Forward (LOCF): The last completed evaluation from the previous visit was carried forward to impute missing data at later visits.
Time Frame: Weeks 2 (first dose of adalimumab in prior phase 3 study), 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, and 216
Population: All participants with evaluable data at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | EW/EW/EW | EW/EOW/EW | EW/PBO/EW
Number analyzed (Participants) | 88 | 90 | 92
percentage of participants
  Week 2: number analyzed (Participants) | 88 | 88 | 91
  Week 2 | 34.1 | 39.8 | 34.1
  Week 4 | 38.6 | 41.1 | 40.2
  Week 8 | 51.1 | 48.9 | 47.8
  Week 12 | 52.3 | 55.6 | 51.1
  Week 16 | 50.0 | 56.7 | 45.7
  Week 20 | 56.8 | 45.6 | 45.7
  Week 24 | 48.9 | 47.8 | 42.4
  Week 36 | 62.5 | 54.4 | 52.2
  Week 48 | 58.0 | 55.6 | 58.7
  Week 60 | 62.5 | 57.8 | 58.7
  Week 72 | 59.1 | 61.1 | 53.3
  Week 84 | 56.8 | 56.7 | 55.4
  Week 96 | 56.8 | 54.4 | 53.3
  Week 108 | 60.2 | 56.7 | 53.3
  Week 120 | 56.8 | 52.2 | 45.7
  Week 132 | 52.3 | 52.2 | 50.0
  Week 144 | 51.1 | 54.4 | 52.2
  Week 156 | 48.9 | 52.2 | 50.0
  Week 168 | 52.3 | 53.3 | 46.7
  Week 180 | 51.1 | 54.4 | 46.7
  Week 192 | 51.1 | 55.6 | 46.7
  Week 204 | 50.0 | 54.4 | 46.7
  Week 216 | 50.0 | 54.4 | 46.7

2. Primary Outcome: Percentage of Participants in the PBO/EW/EW Analysis Population Achieving Clinical Response Per HiSCR at Each Visit
Description: Clinical response per HiSCR defined as percent reduction from baseline of the prior phase 3 study in the abscess and inflammatory nodule ≥ 50% (AN50) with no increase in the abscess count and no increase in the draining fistula count. LOCF: The last completed evaluation from the previous visit was carried forward to impute missing data at later visits.
Time Frame: Entry of Period B in prior phase 3 study, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, and 204
Population: All participants with evaluable data at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | PBO/EW/EW
Number analyzed (Participants) | 115
percentage of participants
  Entry of Period B | 26.1
  Week 12: number analyzed (Participants) | 114
  Week 12 | 54.4
  Week 24: number analyzed (Participants) | 114
  Week 24 | 57.9
  Week 36: number analyzed (Participants) | 114
  Week 36 | 57.0
  Week 48: number analyzed (Participants) | 114
  Week 48 | 60.5
  Week 60: number analyzed (Participants) | 114
  Week 60 | 57.0
  Week 72: number analyzed (Participants) | 114
  Week 72 | 50.0
  Week 84: number analyzed (Participants) | 114
  Week 84 | 50.0
  Week 96: number analyzed (Participants) | 114
  Week 96 | 53.5
  Week 108: number analyzed (Participants) | 114
  Week 108 | 52.6
  Week 120: number analyzed (Participants) | 114
  Week 120 | 53.5
  Week 132: number analyzed (Participants) | 114
  Week 132 | 56.1
  Week 144: number analyzed (Participants) | 114
  Week 144 | 51.8
  Week 156: number analyzed (Participants) | 114
  Week 156 | 52.6
  Week 168: number analyzed (Participants) | 114
  Week 168 | 55.3
  Week 180: number analyzed (Participants) | 114
  Week 180 | 54.4
  Week 192: number analyzed (Participants) | 114
  Week 192 | 53.5
  Week 204: number analyzed (Participants) | 114
  Week 204 | 53.5

3. Primary Outcome: Percentage of Participants in the PBO/PBO/EW Analysis Population Achieving Clinical Response Per HiSCR at Each Visit
Description: as for outcome 2
Time Frame: Entry of M12-555, Weeks 4, 8, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, and 192
Population: All participants with evaluable data at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | PBO/PBO/EW
Number analyzed (Participants) | 123
percentage of participants
  Entry of M12-555 | 19.5
  Week 4: number analyzed (Participants) | 122
  Week 4 | 46.7
  Week 8: number analyzed (Participants) | 122
  Week 8 | 51.6
  Week 12: number analyzed (Participants) | 122
  Week 12 | 48.4
  Week 18: number analyzed (Participants) | 122
  Week 18 | 57.4
  Week 24: number analyzed (Participants) | 122
  Week 24 | 55.7
  Week 36: number analyzed (Participants) | 122
  Week 36 | 60.7
  Week 48: number analyzed (Participants) | 122
  Week 48 | 54.9
  Week 60: number analyzed (Participants) | 122
  Week 60 | 55.7
  Week 72: number analyzed (Participants) | 122
  Week 72 | 54.9
  Week 84: number analyzed (Participants) | 122
  Week 84 | 54.9
  Week 96: number analyzed (Participants) | 122
  Week 96 | 57.4
  Week 108: number analyzed (Participants) | 122
  Week 108 | 54.9
  Week 120: number analyzed (Participants) | 122
  Week 120 | 52.5
  Week 132: number analyzed (Participants) | 122
  Week 132 | 54.1
  Week 144: number analyzed (Participants) | 122
  Week 144 | 51.6
  Week 156: number analyzed (Participants) | 122
  Week 156 | 50.8
  Week 168: number analyzed (Participants) | 122
  Week 168 | 51.6
  Week 180: number analyzed (Participants) | 122
  Week 180 | 51.6
  Week 192: number analyzed (Participants) | 122
  Week 192 | 51.6

4. Primary Outcome: Percentage of Participants in the EW/EW/EW Analysis Population Who Achieved Abscess and Inflammatory Nodule (AN) Count of 0, 1, or 2 at Each Visit
Description: The percentage of participants with AN counts lowered to 0, 1, or 2 at each visit. LOCF: The last completed evaluation from the previous visit was carried forward to impute missing data at later visits.
Time Frame: as for outcome 1
Population: All participants with evaluable data at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | EW/EW/EW
Number analyzed (Participants) | 88
percentage of participants
  Week 2 | 22.7
  Week 4 | 28.4
  Week 8 | 38.6
  Week 12 | 35.2
  Week 16 | 37.5
  Week 20 | 42.0
  Week 24 | 36.4
  Week 36 | 48.9
  Week 48 | 46.6
  Week 60 | 43.2
  Week 72 | 50.0
  Week 84 | 45.5
  Week 96 | 44.3
  Week 108 | 46.6
  Week 120 | 44.3
  Week 132 | 44.3
  Week 144 | 43.2
  Week 156 | 45.5
  Week 168 | 46.6
  Week 180 | 46.6
  Week 192 | 47.7
  Week 204 | 47.7
  Week 216 | 46.6

5. Primary Outcome: Percentage of Participants in the EW/EOW/EW, EW/PBO/EW, and PBO/PBO/EW Analysis Populations Who Achieved AN Count of 0, 1, or 2 at Each Visit
Description: as for outcome 4
Time Frame: Entry of M12-555, Weeks 4, 8, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, and 192
Population: All participants with evaluable data at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | EW/EOW/EW | EW/PBO/EW | PBO/PBO/EW
Number analyzed (Participants) | 90 | 92 | 123
percentage of participants
  Entry of M12-555 | 31.1 | 22.8 | 21.1
  Week 4: number analyzed (Participants) | 87 | 92 | 122
  Week 4 | 35.6 | 34.8 | 44.3
  Week 8: number analyzed (Participants) | 88 | 92 | 122
  Week 8 | 43.2 | 42.4 | 53.3
  Week 12: number analyzed (Participants) | 88 | 92 | 122
  Week 12 | 45.5 | 44.6 | 45.1
  Week 18: number analyzed (Participants) | 88 | 92 | 122
  Week 18 | 50.0 | 41.3 | 50.0
  Week 24: number analyzed (Participants) | 88 | 92 | 122
  Week 24 | 43.2 | 46.7 | 57.4
  Week 36: number analyzed (Participants) | 88 | 92 | 122
  Week 36 | 54.5 | 45.7 | 57.4
  Week 48: number analyzed (Participants) | 88 | 92 | 122
  Week 48 | 50.0 | 42.4 | 52.5
  Week 60: number analyzed (Participants) | 88 | 92 | 122
  Week 60 | 48.9 | 43.5 | 51.6
  Week 72: number analyzed (Participants) | 88 | 92 | 122
  Week 72 | 50.0 | 43.5 | 54.1
  Week 84: number analyzed (Participants) | 88 | 92 | 122
  Week 84 | 53.4 | 44.6 | 50.8
  Week 96: number analyzed (Participants) | 88 | 92 | 122
  Week 96 | 51.1 | 40.2 | 52.5
  Week 108: number analyzed (Participants) | 88 | 92 | 122
  Week 108 | 51.1 | 40.2 | 51.6
  Week 120: number analyzed (Participants) | 88 | 92 | 122
  Week 120 | 46.6 | 37.0 | 52.5
  Week 132: number analyzed (Participants) | 88 | 92 | 122
  Week 132 | 51.1 | 37.0 | 53.3
  Week 144: number analyzed (Participants) | 88 | 92 | 122
  Week 144 | 48.9 | 41.3 | 52.5
  Week 156: number analyzed (Participants) | 88 | 92 | 122
  Week 156 | 47.7 | 39.1 | 51.6
  Week 168: number analyzed (Participants) | 88 | 92 | 122
  Week 168 | 51.1 | 35.9 | 51.6
  Week 180: number analyzed (Participants) | 88 | 92 | 122
  Week 180 | 51.1 | 35.9 | 51.6
  Week 192: number analyzed (Participants) | 88 | 92 | 122
  Week 192 | 51.1 | 35.9 | 51.6

6. Primary Outcome: Percentage of Participants in the PBO/EW/EW Analysis Population Who Achieved AN Count of 0, 1, or 2 at Each Visit
Description: as for outcome 4
Time Frame: as for outcome 2
Population: All participants with evaluable data at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | PBO/EW/EW
Number analyzed (Participants) | 115
percentage of participants
  Entry of Period B | 20.0
  Week 12: number analyzed (Participants) | 114
  Week 12 | 38.6
  Week 24: number analyzed (Participants) | 114
  Week 24 | 43.0
  Week 36: number analyzed (Participants) | 114
  Week 36 | 42.1
  Week 48: number analyzed (Participants) | 114
  Week 48 | 43.9
  Week 60: number analyzed (Participants) | 114
  Week 60 | 45.6
  Week 72: number analyzed (Participants) | 114
  Week 72 | 43.9
  Week 84: number analyzed (Participants) | 114
  Week 84 | 43.9
  Week 96: number analyzed (Participants) | 114
  Week 96 | 46.5
  Week 108: number analyzed (Participants) | 114
  Week 108 | 42.1
  Week 120: number analyzed (Participants) | 114
  Week 120 | 45.6
  Week 132: number analyzed (Participants) | 114
  Week 132 | 46.5
  Week 144: number analyzed (Participants) | 114
  Week 144 | 49.1
  Week 156: number analyzed (Participants) | 114
  Week 156 | 45.6
  Week 168: number analyzed (Participants) | 114
  Week 168 | 46.5
  Week 180: number analyzed (Participants) | 114
  Week 180 | 45.6
  Week 192: number analyzed (Participants) | 114
  Week 192 | 45.6
  Week 204: number analyzed (Participants) | 114
  Week 204 | 45.6

7. Primary Outcome: Modified Sartorius Score: Change From Baseline to Each Visit for Participants in the EW/EW/EW Analysis Population
Description: The Sartorius Scale is used to quantify the severity of HS. Points are awarded for 12 body areas (left and right axillae, left and right sub/inframammary areas, intermammary area, left and right buttocks, left and right inguino-crural folds, perianal area, perineal area, and other): points were awarded for nodules (2 points for each); abscesses (4 points); fistulas (4 points); scars (1 point); other findings (1 point); and longest distance between two lesions (2-6 points, 0 if no lesions); and if lesions are separated by normal skin (yes-0 points; no-6 points). The total Sartorius score is the sum of the 12 regional scores. Higher scores indicate greater severity of HS. A negative change indicates decrease in severity. LOCF: The last completed evaluation from the previous visit was carried forward to impute missing data at later visits.
Time Frame: Baseline (in prior phase 3 study) to Weeks 2 (first dose of adalimumab in prior phase 3 study), 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, and 216
Population: All participants with evaluable data at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EW/EW/EW
Number analyzed (Participants) | 88
units on a scale
  Week 2 | -18.0 (25.27)
  Week 4 | -21.0 (31.81)
  Week 8 | -22.8 (35.45)
  Week 12 | -23.9 (48.30)
  Week 16 | -26.6 (54.63)
  Week 20 | -32.1 (73.69)
  Week 24 | -36.6 (74.99)
  Week 36 | -41.6 (93.11)
  Week 48 | -42.2 (115.22)
  Week 60 | -41.9 (119.98)
  Week 72 | -43.2 (122.30)
  Week 84 | -42.8 (123.18)
  Week 96 | -43.2 (126.21)
  Week 108 | -43.2 (124.92)
  Week 120 | -43.4 (127.65)
  Week 132 | -42.5 (128.45)
  Week 144 | -42.4 (129.37)
  Week 156 | -40.7 (130.30)
  Week 168 | -41.5 (130.40)
  Week 180 | -41.8 (129.89)
  Week 192 | -41.9 (130.46)
  Week 204 | -41.4 (130.72)
  Week 216 | -41.4 (130.94)

8. Primary Outcome: Modified Sartorius Score: Change From Baseline to Each Visit for Participants in the EW/EOW/EW, EW/PBO/EW, and PBO/PBO/EW Analysis Populations
Description: as for outcome 7
Time Frame: Baseline (in prior phase 3 study) to Entry of M12-555 and Weeks 4, 8, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, and 192
Population: All participants with evaluable data at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EW/EOW/EW | EW/PBO/EW | PBO/PBO/EW
Number analyzed (Participants) | 90 | 92 | 123
units on a scale
  Entry of M12-555 | -23.1 (56.94) | -10.5 (56.74) | 0.2 (51.35)
  Week 4: number analyzed (Participants) | 87 | 92 | 122
  Week 4 | -30.2 (48.99) | -18.8 (56.52) | -16.2 (56.16)
  Week 8: number analyzed (Participants) | 88 | 92 | 122
  Week 8 | -34.9 (47.42) | -21.2 (63.26) | -24.8 (51.55)
  Week 12: number analyzed (Participants) | 88 | 92 | 122
  Week 12 | -34.8 (55.71) | -25.5 (57.92) | -26.2 (54.58)
  Week 18: number analyzed (Participants) | 88 | 92 | 122
  Week 18 | -35.9 (47.92) | -26.2 (60.59) | -32.3 (48.60)
  Week 24: number analyzed (Participants) | 88 | 92 | 122
  Week 24 | -37.1 (47.39) | -24.1 (61.52) | -33.5 (50.20)
  Week 36: number analyzed (Participants) | 88 | 92 | 122
  Week 36 | -37.1 (46.07) | -24.7 (63.81) | -33.6 (57.58)
  Week 48: number analyzed (Participants) | 88 | 92 | 122
  Week 48 | -37.5 (47.94) | -24.8 (63.21) | -30.2 (64.84)
  Week 60: number analyzed (Participants) | 88 | 92 | 122
  Week 60 | -34.8 (50.17) | -22.6 (65.06) | -31.7 (66.33)
  Week 72: number analyzed (Participants) | 88 | 92 | 122
  Week 72 | -35.4 (55.22) | -20.1 (64.52) | -31.8 (65.26)
  Week 84: number analyzed (Participants) | 88 | 92 | 122
  Week 84 | -36.6 (51.33) | -20.0 (66.02) | -29.5 (65.79)
  Week 96: number analyzed (Participants) | 88 | 92 | 122
  Week 96 | -34.0 (49.42) | -18.3 (65.14) | -29.0 (68.85)
  Week 108: number analyzed (Participants) | 88 | 92 | 122
  Week 108 | -34.0 (54.41) | -18.3 (66.88) | -28.4 (71.52)
  Week 120: number analyzed (Participants) | 88 | 92 | 122
  Week 120 | -31.8 (60.85) | -16.2 (66.82) | -28.3 (70.37)
  Week 132: number analyzed (Participants) | 88 | 92 | 122
  Week 132 | -35.1 (53.01) | -16.7 (66.87) | -28.8 (69.79)
  Week 144: number analyzed (Participants) | 88 | 92 | 122
  Week 144 | -35.1 (53.94) | -16.6 (67.30) | -28.6 (70.03)
  Week 156: number analyzed (Participants) | 88 | 92 | 122
  Week 156 | -34.7 (53.95) | -15.7 (67.09) | -28.0 (69.11)
  Week 168: number analyzed (Participants) | 88 | 92 | 122
  Week 168 | -35.6 (53.72) | -15.5 (67.40) | -28.7 (69.81)
  Week 180: number analyzed (Participants) | 88 | 92 | 122
  Week 180 | -35.6 (53.64) | -15.4 (67.39) | -28.7 (69.81)
  Week 192: number analyzed (Participants) | 88 | 92 | 122
  Week 192 | -35.6 (53.64) | -15.4 (67.39) | -28.7 (69.81)

9. Primary Outcome: Modified Sartorius Score: Change From Baseline to Each Visit for Participants in the PBO/EW/EW Analysis Population
Description: as for outcome 7
Time Frame: Baseline (in prior phase 3 study) to Entry of Period B in prior phase 3 study and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, and 204
Population: All participants with evaluable data at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PBO/EW/EW
Number analyzed (Participants) | 115
units on a scale
  Entry of Period B | -18.0 (38.32)
  Week 12: number analyzed (Participants) | 114
  Week 12 | -43.2 (48.07)
  Week 24: number analyzed (Participants) | 114
  Week 24 | -43.0 (53.08)
  Week 36: number analyzed (Participants) | 114
  Week 36 | -49.5 (57.05)
  Week 48: number analyzed (Participants) | 114
  Week 48 | -47.1 (61.95)
  Week 60: number analyzed (Participants) | 114
  Week 60 | -46.2 (60.94)
  Week 72: number analyzed (Participants) | 114
  Week 72 | -44.5 (67.13)
  Week 84: number analyzed (Participants) | 114
  Week 84 | -46.8 (64.57)
  Week 96: number analyzed (Participants) | 114
  Week 96 | -45.5 (70.63)
  Week 108: number analyzed (Participants) | 114
  Week 108 | -45.0 (74.15)
  Week 120: number analyzed (Participants) | 114
  Week 120 | -45.9 (75.30)
  Week 132: number analyzed (Participants) | 114
  Week 132 | -44.4 (78.09)
  Week 144: number analyzed (Participants) | 114
  Week 144 | -45.4 (76.53)
  Week 156: number analyzed (Participants) | 114
  Week 156 | -46.0 (76.17)
  Week 168: number analyzed (Participants) | 114
  Week 168 | -46.1 (75.84)
  Week 180: number analyzed (Participants) | 114
  Week 180 | -45.8 (75.96)
  Week 192: number analyzed (Participants) | 114
  Week 192 | -45.8 (75.89)
  Week 204: number analyzed (Participants) | 114
  Week 204 | -45.9 (75.96)

10. Primary Outcome: Percentage of Participants in the EW/EW/EW Analysis Population Achieving Skin Pain NRS30 - At Worst at Each Visit Among Participants With Baseline Skin Pain NRS At Worst ≥ 3
Description: The Patient's Global Assessment of Skin Pain Numeric Rating Scale (NRS) was used to assess the worst skin pain and the average skin pain due to HS. Ratings for the 2 items range from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). The assessments were completed on a daily diary by participants before they went to bed and responded to the items based on a recall period of the "last 24 hours." The percentage of participants who achieved at least 30% reduction and at least 1 unit reduction from Baseline in the Patient's Global Assessment of Skin Pain (NRS30) - at worst at each visit among participants with baseline skin pain NRS - at worst ≥ 3 are presented. Weekly averages of daily assessments were analyzed. LOCF: The last completed evaluation from the previous visit was carried forward to impute missing data at later visits.
Time Frame: Weeks 2 (first dose of adalimumab in prior phase 3 study), 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, and 192
Population: All participants with baseline skin pain NRS-at worst ≥3 and with evaluable data at given time point
Measure: Number; unit: percentage of participants
Arm/Group | EW/EW/EW
Number analyzed (Participants) | 63
percentage of participants
  Week 2 | 47.6
  Week 4 | 46.0
  Week 8 | 44.4
  Week 12 | 42.9
  Week 16 | 46.0
  Week 20 | 50.8
  Week 24 | 54.0
  Week 36 | 58.7
  Week 48 | 54.0
  Week 60 | 52.4
  Week 72 | 54.0
  Week 84 | 52.4
  Week 96 | 49.2
  Week 108 | 54.0
  Week 120 | 50.8
  Week 132 | 46.0
  Week 144 | 54.0
  Week 156 | 52.4
  Week 168 | 52.4
  Week 180 | 52.4
  Week 192 | 52.4

11. Primary Outcome: Percentage of Participants in the EW/EOW/EW, EW/PBO/EW, and PBO/PBO/EW Analysis Populations Achieving Skin Pain NRS30 - At Worst at Each Visit Among Participants With Baseline Skin Pain NRS At Worst ≥ 3
Description: The NRS was used to assess the worst skin pain and the average skin pain due to HS. Ratings for the 2 items range from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). The assessments were completed on a daily diary by participants before they went to bed and responded to the items based on a recall period of the "last 24 hours." The percentage of participants who achieved at least 30% reduction and at least 1 unit reduction from Baseline in the NRS (NRS30) - at worst at each visit among participants with baseline skin pain NRS - at worst ≥ 3 are presented. Weekly averages of daily assessments were analyzed. LOCF: The last completed evaluation from the previous visit was carried forward to impute missing data at later visits.
Time Frame: Entry of M12-555, and Weeks 4, 8, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, and 192
Population: All participants with baseline skin pain NRS-at worst ≥3 and with evaluable data at given time point
Measure: Number; unit: percentage of participants
Arm/Group | EW/EOW/EW | EW/PBO/EW | PBO/PBO/EW
Number analyzed (Participants) | 65 | 64 | 84
percentage of participants
  Entry of M12-555 | 40.0 | 21.9 | 22.6
  Week 4: number analyzed (Participants) | 61 | 58 | 83
  Week 4 | 47.5 | 43.1 | 44.6
  Week 8: number analyzed (Participants) | 62 | 63 | 83
  Week 8 | 45.2 | 47.6 | 51.8
  Week 12: number analyzed (Participants) | 63 | 63 | 83
  Week 12 | 41.3 | 54.0 | 51.8
  Week 18: number analyzed (Participants) | 63 | 63 | 83
  Week 18 | 47.6 | 50.8 | 55.4
  Week 24: number analyzed (Participants) | 63 | 63 | 83
  Week 24 | 42.9 | 47.6 | 54.2
  Week 36: number analyzed (Participants) | 63 | 63 | 83
  Week 36 | 49.2 | 47.6 | 55.4
  Week 48: number analyzed (Participants) | 63 | 63 | 83
  Week 48 | 47.6 | 50.8 | 56.6
  Week 60: number analyzed (Participants) | 63 | 63 | 83
  Week 60 | 47.6 | 50.8 | 50.6
  Week 72: number analyzed (Participants) | 63 | 63 | 83
  Week 72 | 47.6 | 42.9 | 50.6
  Week 84: number analyzed (Participants) | 63 | 63 | 83
  Week 84 | 50.8 | 46.0 | 48.2
  Week 96: number analyzed (Participants) | 63 | 63 | 83
  Week 96 | 50.8 | 55.6 | 48.2
  Week 108: number analyzed (Participants) | 63 | 63 | 83
  Week 108 | 50.8 | 42.9 | 50.6
  Week 120: number analyzed (Participants) | 63 | 63 | 83
  Week 120 | 42.9 | 47.6 | 45.8
  Week 132: number analyzed (Participants) | 63 | 63 | 83
  Week 132 | 41.3 | 47.6 | 48.2
  Week 144: number analyzed (Participants) | 63 | 63 | 83
  Week 144 | 41.3 | 50.8 | 47.0
  Week 156: number analyzed (Participants) | 63 | 63 | 83
  Week 156 | 39.7 | 46.0 | 49.4
  Week 168: number analyzed (Participants) | 63 | 63 | 83
  Week 168 | 41.3 | 49.2 | 48.2
  Week 180: number analyzed (Participants) | 63 | 63 | 83
  Week 180 | 41.3 | 49.2 | 48.2
  Week 192: number analyzed (Participants) | 63 | 63 | 83
  Week 192 | 41.3 | 49.2 | 48.2

12. Primary Outcome: Percentage of Participants in the PBO/EW/EW Analysis Population Achieving Skin Pain NRS30 - At Worst at Each Visit Among Participants With Baseline Skin Pain NRS At Worst ≥ 3
Description: as for outcome 11
Time Frame: as for outcome 2
Population: All participants with baseline skin pain NRS-at worst ≥3 and with evaluable data at given time point
Measure: Number; unit: percentage of participants
Arm/Group | PBO/EW/EW
Number analyzed (Participants) | 79
percentage of participants
  Entry of Period B | 31.6
  Week 12: number analyzed (Participants) | 64
  Week 12 | 51.6
  Week 24: number analyzed (Participants) | 76
  Week 24 | 55.3
  Week 36: number analyzed (Participants) | 77
  Week 36 | 55.8
  Week 48: number analyzed (Participants) | 77
  Week 48 | 53.2
  Week 60: number analyzed (Participants) | 77
  Week 60 | 58.4
  Week 72: number analyzed (Participants) | 77
  Week 72 | 64.9
  Week 84: number analyzed (Participants) | 77
  Week 84 | 63.6
  Week 96: number analyzed (Participants) | 77
  Week 96 | 62.3
  Week 108: number analyzed (Participants) | 78
  Week 108 | 55.1
  Week 120: number analyzed (Participants) | 78
  Week 120 | 56.4
  Week 132: number analyzed (Participants) | 78
  Week 132 | 53.8
  Week 144: number analyzed (Participants) | 78
  Week 144 | 55.1
  Week 156: number analyzed (Participants) | 78
  Week 156 | 51.3
  Week 168: number analyzed (Participants) | 78
  Week 168 | 57.7
  Week 180: number analyzed (Participants) | 78
  Week 180 | 57.7
  Week 192: number analyzed (Participants) | 78
  Week 192 | 56.4
  Week 204: number analyzed (Participants) | 78
  Week 204 | 57.7

13. Primary Outcome: Percentage of Participants in the EW/EW/EW Analysis Population Achieving Skin Pain NRS30 - On Average at Each Visit Among Participants With Baseline Skin Pain NRS On Average ≥ 3
Description: The NRS was used to assess the worst skin pain and the average skin pain due to HS. Ratings for the 2 items range from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). The assessments were completed on a daily diary by participants before they went to bed and responded to the items based on a recall period of the "last 24 hours." The percentage of participants who achieved at least 30% reduction and at least 1 unit reduction from Baseline in the NRS (NRS30) - on average at each visit among participants with baseline skin pain NRS - on average ≥ 3 are presented. Weekly averages of daily assessments were analyzed. LOCF: The last completed evaluation from the previous visit was carried forward to impute missing data at later visits.
Time Frame: as for outcome 10
Population: All participants with baseline skin pain NRS - on average ≥ 3 and with evaluable data at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | EW/EW/EW
Number analyzed (Participants) | 50
percentage of participants
  Week 2 | 56.0
  Week 4 | 52.0
  Week 8 | 48.0
  Week 12 | 46.0
  Week 16 | 40.0
  Week 20 | 50.0
  Week 24 | 46.0
  Week 36 | 58.0
  Week 48 | 56.0
  Week 60 | 56.0
  Week 72 | 56.0
  Week 84 | 56.0
  Week 96 | 54.0
  Week 108 | 50.0
  Week 120 | 48.0
  Week 132 | 56.0
  Week 144 | 56.0
  Week 156 | 58.0
  Week 168 | 56.0
  Week 180 | 56.0
  Week 192 | 56.0

14. Primary Outcome: Percentage of Participants in the EW/EOW/EW, EW/PBO/EW, and PBO/PBO/EW Analysis Populations Achieving Skin Pain NRS30 - On Average at Each Visit Among Participants With Baseline Skin Pain NRS On Average ≥ 3
Description: as for outcome 13
Time Frame: Entry of M12-555, and Weeks 4, 8, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, and 192
Population: All participants with baseline skin pain NRS - on average ≥ 3 and with evaluable data at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | EW/EOW/EW | EW/PBO/EW | PBO/PBO/EW
Number analyzed (Participants) | 55 | 53 | 69
percentage of participants
  Entry of M12-555 | 43.6 | 37.7 | 31.9
  Week 4: number analyzed (Participants) | 51 | 47 | 68
  Week 4 | 49.0 | 46.8 | 61.8
  Week 8: number analyzed (Participants) | 52 | 52 | 68
  Week 8 | 46.2 | 55.8 | 61.8
  Week 12: number analyzed (Participants) | 53 | 52 | 68
  Week 12 | 39.6 | 59.6 | 58.8
  Week 18: number analyzed (Participants) | 53 | 52 | 68
  Week 18 | 45.3 | 59.6 | 63.2
  Week 24: number analyzed (Participants) | 53 | 52 | 68
  Week 24 | 39.6 | 53.8 | 54.4
  Week 36: number analyzed (Participants) | 53 | 52 | 68
  Week 36 | 45.3 | 48.1 | 58.8
  Week 48: number analyzed (Participants) | 53 | 52 | 68
  Week 48 | 47.2 | 51.9 | 58.8
  Week 60: number analyzed (Participants) | 53 | 52 | 68
  Week 60 | 43.4 | 53.8 | 55.9
  Week 72: number analyzed (Participants) | 53 | 52 | 68
  Week 72 | 47.2 | 59.6 | 55.9
  Week 84: number analyzed (Participants) | 53 | 52 | 68
  Week 84 | 49.1 | 48.1 | 52.9
  Week 96: number analyzed (Participants) | 53 | 52 | 68
  Week 96 | 47.2 | 57.7 | 57.4
  Week 108: number analyzed (Participants) | 53 | 52 | 68
  Week 108 | 49.1 | 44.2 | 54.4
  Week 120: number analyzed (Participants) | 53 | 52 | 68
  Week 120 | 39.6 | 48.1 | 54.4
  Week 132: number analyzed (Participants) | 53 | 52 | 68
  Week 132 | 43.4 | 50.0 | 54.4
  Week 144: number analyzed (Participants) | 53 | 52 | 68
  Week 144 | 43.4 | 50.0 | 54.4
  Week 156: number analyzed (Participants) | 53 | 52 | 68
  Week 156 | 43.4 | 46.2 | 55.9
  Week 168: number analyzed (Participants) | 53 | 52 | 68
  Week 168 | 43.4 | 48.1 | 54.4
  Week 180: number analyzed (Participants) | 53 | 52 | 68
  Week 180 | 43.4 | 48.1 | 54.4
  Week 192: number analyzed (Participants) | 53 | 52 | 68
  Week 192 | 43.4 | 48.1 | 54.4

15. Primary Outcome: Percentage of Participants in the PBO/EW/EW Analysis Population Achieving Skin Pain NRS30 - On Average at Each Visit Among Participants With Baseline Skin Pain NRS On Average ≥ 3
Description: as for outcome 13
Time Frame: as for outcome 2
Population: All participants with baseline skin pain NRS - on average ≥ 3 and with evaluable data at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | PBO/EW/EW
Number analyzed (Participants) | 62
percentage of participants
  Entry of Period B | 30.6
  Week 12: number analyzed (Participants) | 49
  Week 12 | 59.2
  Week 24: number analyzed (Participants) | 59
  Week 24 | 61.0
  Week 36: number analyzed (Participants) | 60
  Week 36 | 61.7
  Week 48: number analyzed (Participants) | 60
  Week 48 | 53.3
  Week 60: number analyzed (Participants) | 60
  Week 60 | 60.0
  Week 72: number analyzed (Participants) | 60
  Week 72 | 58.3
  Week 84: number analyzed (Participants) | 60
  Week 84 | 60.0
  Week 96: number analyzed (Participants) | 60
  Week 96 | 61.7
  Week 108: number analyzed (Participants) | 61
  Week 108 | 62.3
  Week 120: number analyzed (Participants) | 61
  Week 120 | 62.3
  Week 132: number analyzed (Participants) | 61
  Week 132 | 59.0
  Week 144: number analyzed (Participants) | 61
  Week 144 | 60.7
  Week 156: number analyzed (Participants) | 61
  Week 156 | 55.7
  Week 168: number analyzed (Participants) | 61
  Week 168 | 62.3
  Week 180: number analyzed (Participants) | 61
  Week 180 | 62.3
  Week 192: number analyzed (Participants) | 61
  Week 192 | 60.7
  Week 204: number analyzed (Participants) | 61
  Week 204 | 62.3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 70 days after the last dose of study drug (up to 225 weeks).
Description: TEAEs and TESAEs were defined as AEs and SAEs with an onset date on or after the first dose of adalimumab in either M12-555 or in prior studies M11-313 or M11-810, excluding AEs and SAEs with onset date during a protocol-defined treatment gap.
Groups:
- All Adalimumab: Participants who received at least 1 dose of adalimumab (40 mg every week) in M12-555.
Arm/Group | All Adalimumab
Serious Adverse Events (participants affected / at risk) | 99/508
Other Adverse Events (participants affected / at risk) | 349/508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Adalimumab (N=508)
LYMPHADENITIS (Blood and lymphatic system disorders) | 1
ANGINA PECTORIS (Cardiac disorders) | 2
CARDIAC ARREST (Cardiac disorders) | 1
CARDIAC FAILURE (Cardiac disorders) | 1
PALPITATIONS (Cardiac disorders) | 2
ODONTOGENIC CYST (Congenital, familial and genetic disorders) | 1
AUTOIMMUNE PANCREATITIS (Gastrointestinal disorders) | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 1
INCARCERATED UMBILICAL HERNIA (Gastrointestinal disorders) | 1
PERITONEAL CYST (Gastrointestinal disorders) | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1
PYREXIA (General disorders) | 1
CHOLANGITIS (Hepatobiliary disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 2
APPENDICITIS (Infections and infestations) | 2
CELLULITIS (Infections and infestations) | 2
ERYSIPELAS (Infections and infestations) | 1
GROIN ABSCESS (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
PERITONITIS (Infections and infestations) | 1
PERITONSILLAR ABSCESS (Infections and infestations) | 1
PERIUMBILICAL ABSCESS (Infections and infestations) | 1
PILONIDAL CYST (Infections and infestations) | 2
PNEUMONIA (Infections and infestations) | 3
PNEUMONIA CHLAMYDIAL (Infections and infestations) | 1
PNEUMONIA VIRAL (Infections and infestations) | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2
PYELONEPHRITIS (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 2
SEPTIC SHOCK (Infections and infestations) | 2
VULVAL ABSCESS (Infections and infestations) | 1
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 1
CONTUSION (Injury, poisoning and procedural complications) | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
MENISCUS INJURY (Injury, poisoning and procedural complications) | 1
PROCEDURAL DIZZINESS (Injury, poisoning and procedural complications) | 1
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1
RADIAL HEAD DISLOCATION (Injury, poisoning and procedural complications) | 1
SCAR (Injury, poisoning and procedural complications) | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
AUTOANTIBODY POSITIVE (Investigations) | 1
BODY TEMPERATURE INCREASED (Investigations) | 1
OBESITY (Metabolism and nutrition disorders) | 3
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2
JOINT INSTABILITY (Musculoskeletal and connective tissue disorders) | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1
BREAST CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CARDIAC MYXOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
INVASIVE BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PAPILLARY CYSTADENOMA LYMPHOMATOSUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SEMINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
COMA HEPATIC (Nervous system disorders) | 1
HEMIPLEGIA (Nervous system disorders) | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1
SUICIDAL IDEATION (Psychiatric disorders) | 2
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2
URETERIC OBSTRUCTION (Renal and urinary disorders) | 1
DYSFUNCTIONAL UTERINE BLEEDING (Reproductive system and breast disorders) | 1
OVARIAN CYST (Reproductive system and breast disorders) | 1
PELVIC PROLAPSE (Reproductive system and breast disorders) | 1
UTERINE CYST (Reproductive system and breast disorders) | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
CUTIS LAXA (Skin and subcutaneous tissue disorders) | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 29
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 1
PYODERMA GANGRENOSUM (Skin and subcutaneous tissue disorders) | 1
SEXUAL ABUSE (Social circumstances) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
HYPERTENSION (Vascular disorders) | 2
HYPERTENSIVE CRISIS (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Adalimumab (N=508)
DIARRHOEA (Gastrointestinal disorders) | 33
NAUSEA (Gastrointestinal disorders) | 32
PYREXIA (General disorders) | 29
BRONCHITIS (Infections and infestations) | 37
GASTROENTERITIS (Infections and infestations) | 26
INFLUENZA (Infections and infestations) | 40
NASOPHARYNGITIS (Infections and infestations) | 92
SINUSITIS (Infections and infestations) | 29
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 84
URINARY TRACT INFECTION (Infections and infestations) | 40
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 38
BACK PAIN (Musculoskeletal and connective tissue disorders) | 33
HEADACHE (Nervous system disorders) | 80
COUGH (Respiratory, thoracic and mediastinal disorders) | 27
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 125
HYPERTENSION (Vascular disorders) | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.